CLINICAL TRIAL: NCT04514835
Title: A Phase Ⅱ Trials of Sintilimab as Consolidation Therapy After Radical Concurrent Chemoradiotherapy in Locally Advanced Unresectable ESCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Feng Wang, DOCTOR, The First Affiliated Hospital of Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IBI308-01
Record Dates: First submitted 2020-08-05; First posted 2020-08-17 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cisplatin+Capecitabine+Sintilimab (Experimental): Cisplatin+Capecitabine+Sintilimab
  Interventions: Drug: Cisplatin+Capecitabine+Sintilimab

INTERVENTIONS:
Drug: Cisplatin+Capecitabine+Sintilimab — The first stage:concurrent chemoradiotherapy，cisplatin，25-30mg/m2 ivgtt d1;capecitabine,800mg/m2, bid d1-5，qw，5weeks;concurrent radiotherapy,1.8-2Gy/d，5d/W，50-50.4Gy.
  second stage:Sintilimab, 200mg,q3w, a total of 3 times，Each infusion lasted for 30-60 min until disease progression or intolerable toxicity, with a maximum duration of no more than 12 months.

SUMMARY:
The purpose of this study is to observe and evaluate the efficacy and safety of Sintilimab for Consolidation Therapy After Radical Concurrent Chemoradiotherapy for Locally Advanced Unresectable Esophageal Squamous Cell Carcinoma

DETAILED DESCRIPTION:
In China, the incidence of esophageal cancer has declined in recent years, but the mortality rate has been ranked fourth. Morbidity and mortality were ranked sixth and fourth in all malignancies, respectively. Therefore, esophageal cancer has always been a major malignant tumor that threatens the health of our residents.We designed a single-arm, open-label, phase II trial of Sintilimab for consolidation therapy after radical concurrent chemoradiotherapylocally advanced esophageal squamous cell carcinoma.The purpose of this study is to observe and evaluate the efficacy and safety of Sintilimab for consolidation therapy after radical concurrent chemoradiotherapy for locally advanced unresectable esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old, both men and women; 2. Histology confirmed as esophageal squamous cell carcinoma; 3. T1bN+M0, T2-T4aN0-2M0 locally advanced stage； 4. Tissue samples should be provided for biomarker analysis, and the newly obtained tissues should be selected. Patients who cannot provide newly obtained tissues can provide 5-8. pieces of 5-um thick paraffin sections; 5. ECOG: 0~1; 6. Expected survival period ≥ 12 weeks; 7. The main organs function normally, that is, the following criteria are met:

1. Blood routine examination:

   1. HB≥90g/L;
   2. ANC ≥ 1.5 × 109 / L;
   3. PLT ≥ 80 × 109 / L;
2. Biochemical examination:

   1. ALB ≥ 30g / L;b.ALT and AST ≤ 2.5ULN; if there is liver metastasis, ALT and AST ≤ 5ULN;c.TBIL ≤ 1.5ULN;d.plasma Cr ≤ 1.5ULN or creatinine clearance (CCr) ≥ 60ml / min; 8.Doppler ultrasound assessment: left ventricular ejection fraction (LVEF) ≥ normal low limit (50%); 9. Women of childbearing age should agree to use contraceptives (such as intrauterine devices, contraceptives or condoms) during the study period and within 6 months after the end of the study; negative serum or urine pregnancy test within 7 days prior to study enrollment And must be non-lactating patients; males should agree to patients who must use contraception during the study period and within 6 months after the end of the study period; 10. Subjects voluntarily joined the study, signed informed consent, and were well-adhered to follow-up.

Exclusion Criteria:

1. Does not meet the above inclusion criteria;
2. Those who are allergic to or sensitive to capecitabine and cisplatin or metabolic disorders;
3. The patient has any active autoimmune disease or a history of autoimmune disease (such as the following, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis,Hyperthyroidism; patients with vitiligo ; Asthma has been completely relieved in childhood, and patients who do not need any intervention after adulthood can be included; asthma patients who require bronchodilators for medical intervention cannot be included);
4. The patient is using immunosuppressive agents or systemic hormonal therapy for immunosuppressive purposes (dose> 10 mg/day of prednisone or other therapeutic hormones) and continues to be used for 2 weeks prior to enrollment;
5. contraindications to radiotherapy;
6. Patients with any severe and/or uncontrolled diseases:Patients with unsatisfactory blood pressure control (systolic blood pressure ≥150mmHg or diastolic blood pressure ≥100 mmHg); myocardial ischemia or myocardial infarction with grade I or above, arrhythmia (including QT interval ≥ 480ms) and grade I cardiac insufficiency;
7. Active or uncontrolled serious infections;
8. Liver diseases such as decompensated liver disease, active hepatitis B (HBV-DNA ≥ 104 copies/ml or 2000 IU/ml) or hepatitis C (positive hepatitis C antibody, and HCV-RNA is higher than the lower limit of detection of the analytical method);
9. Urine routine indicates that urine protein ≥ ++, and confirmed 24-hour urine protein quantitation> 1.0g;
10. The patients whose imaging showed that the tumor had invaded the important vessels or the tumor was likely to invade the important vessels and cause fatal hemorrhage during the follow-up study;
11. Pregnant or lactating women;
12. Patients with other malignancies within 5 years (except for basal cell carcinoma and cervical carcinoma in situ) that have been cured;
13. Patients with a history of psychotropic substance abuse who are unable to quit or have a mental disorder;
14. Patients who have participated in other drug clinical trials within four weeks;
15. At the discretion of the investigator, there are patients with serious concomitant disease that compromises patient safety or affects the patient's completion of the study;
16. The investigator believes that it is not suitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-01-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival（PFS） | up to 1 year
  Evaluation of anti-PD-1 antibody Sintilimab for progression-free survival in patients with locally advanced unresectable esophageal squamous cell carcinoma who did not develop disease after radical concurrent chemoradiotherapy

SECONDARY OUTCOMES:
Objective Response Rate，ORR | At time of surgery
  To evaluate the objective response rate (objective response rate, ORR) of Sintilimab in patients with locally advanced esophageal squamous cell carcinoma who have not progressed after concurrent radiotherapy and chemotherapy

OTHER OUTCOMES:
Overall survival, OS | At time of surgery
  From date of randomization until the date of death from any cause
Exploratory analysis of biomarkers for predicting efficacy | At time of surgery
  The relationship between PD-L1 dynamic expression, ctDNA sequencing and therapeutic effect was evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Feng Wang, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, China